CLINICAL TRIAL: NCT00396084
Title: Randomized, Open Label, Multiple Dose Phase I Study of the Early Bactericidal Activity of Linezolid, Gatifloxacin, Levofloxacin, and Moxifloxacin in HIV-non-infected Adults With Initial Episodes of Sputum Smear-Positive Pulmonary Tuberculosis
Brief Title: Early Bactericidal Activity of Linezolid, Gatifloxacin, Levofloxacin, Isoniazid (INH) and Moxifloxacin in HIV Negative Adults With Initial Episodes of Sputum Smear-Positive Pulmonary Tuberculosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-553
Record Dates: First submitted 2006-11-03; First posted 2006-11-06 (Estimated); Results first posted 2009-06-25 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2010-03-10

CONDITIONS: Tuberculosis
Keywords: Brazil; gatifloxacin; isoniazid; levofloxacin; linezolid; moxifloxacin; tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Gatifloxacin; Isoniazid; Levofloxacin; Linezolid; Moxifloxacin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Gatifloxacin (Experimental): 10 subjects to receive gatifloxacin 400 mg orally once daily for 7 days.
  Interventions: Drug: Gatifloxacin
- Isoniazid (Active Comparator): 20 subjects to receive isoniazid 300 mg orally once daily for 7days.
  Interventions: Drug: Isoniazid
- Levofloxacin (Experimental): 10 subjects to receive levofloxacin 1000 mg orally once daily for 7days.
  Interventions: Drug: Levofloxacin
- Linezolid every 12 hours (Experimental): 10 subjects to receive linezolid 600 mg orally every 12 hours daily for 7 days.
  Interventions: Drug: Linezolid
- Linezolid once daily (Experimental): 10 subjects to receive linezolid 600 mg orally once daily for 7days.
  Interventions: Drug: Linezolid
- Moxifloxacin (Experimental): 10 subjects to receive moxifloxacin 400 mg orally once daily for 7 days.
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Gatifloxacin — Gatifloxacin 400 mg/day x 7 days.
  Arms: Gatifloxacin
Drug: Isoniazid — Isoniazid 300 mg/day x 7 days.
  Arms: Isoniazid
Drug: Levofloxacin — Levofloxacin 1000 mg/day x 7 days.
  Arms: Levofloxacin
Drug: Linezolid — Linezolid 600 mg/day x 7 days; Linezolid 600 mg every 12 hours x 7 days.
  Arms: Linezolid every 12 hours; Linezolid once daily
Drug: Moxifloxacin — Moxifloxacin 400 mg/day x 7 days.
  Arms: Moxifloxacin

SUMMARY:
This study will evaluate the ability of 4 antibiotics to kill the bacteria that cause tuberculosis (TB). The antibiotics to be studied are linezolid, gatifloxacin, levofloxacin, and moxifloxacin. All are approved by the Brazilian health authorities to treat infections caused by germs other than TB. Seventy human immunodeficiency virus (HIV)-negative adults, aged 18-65 years, who have been newly diagnosed with pulmonary (lung) TB, will participate in this study. Study volunteers will be given one of the 4 study drugs or a comparison antibiotic, Isoniazid, which has been used around the world as a standard of care treatment for TB. Volunteers will stay in the hospital for 10 days and be given a study antibiotic 7 of those days. Blood and saliva samples will be taken. Six weeks later, volunteers will return for a final health check. All volunteers will receive 6 months of standard tuberculosis treatment.

DETAILED DESCRIPTION:
Multi-drug resistant tuberculosis now affects all regions of the world and is a significant concern for national tuberculosis (TB) control programs. The development and testing of new drugs and new classes of drugs and immunotherapeutic agents are vital elements in the global response to this challenge. The fluoroquinolones and oxazolidinones represent two promising classes of drugs that show activity against Mycobacterium tuberculosis (MTB). This study is a randomized, open label, multiple dose phase I clinical trial to evaluate the early bactericidal activity (EBA) of gatifloxacin, levofloxacin, moxifloxacin, and linezolid compared with an isoniazid (INH) control arm in patients with newly-diagnosed sputum smear-positive pulmonary tuberculosis (TB). Secondary study objectives are to: compare results of sputum MTB messenger ribonucleic acid (mRNA) clearance with results of a standard EBA study [change in sputum viable counts [colony forming units (CFU)]; compare the rate of clearance of sputum cytokine proteins with results of a standard EBA assay CFU; determine the pharmacokinetics (PK) of the study drugs in patients with smear-positive pulmonary TB; and demonstrate that lack of EBA activity is not due to low serum drug concentrations. Seventy human immunodeficiency virus (HIV) negative adults, aged 18-65 years, who have been newly diagnosed with pulmonary TB, will be enrolled and admitted to the Centro de Pesquisa (Clinical Research Ward) at the Hospital Universitario Cassiano Antonio de Moraes of the Universidade Federal do Espírito Santo in Vitória. The subjects will be randomized to receive gatifloxacin, levofloxacin, moxifloxacin, or INH (control), and after these arms are enrolled, they will be randomized to receive either linezolid (600 mg once daily) or linezolid (600 mg twice daily) or INH (control). During the inpatient stay, study drugs will be given for 7 days following a 2-day drug-free period when baseline sputum bacillary counts will be measured. The 7-day duration of the study drug phase will allow measurement of sputum bactericidal activity both during the first 2 days of study drug administration and between days 2 and 7 of study drug administration to gain additional information on the possible sterilizing activity of the drugs. The extended nature of these EBA studies will allow assessment of this possibility in the study drugs that would be missed if a shorter EBA study was performed. Sputum specimens will be collected for 2 days prior to initiation of study drug in order to establish a baseline quantitative culture result and then specimens will be collected daily thereafter. Sputum specimens will be processed to evaluate changes in mycobacterial mRNA/proteins and cytokine proteins. PK studies will be performed after 5 days of study drug administration (Day 5). Safety evaluations including clinical examination, complete blood counts, and serum total bilirubin, aspartate aminotransferase (AST), creatinine, and urinalysis will be followed to monitor for drug toxicity. Drug susceptibility testing will be performed on an initial sputum isolate and will be repeated after completion of 7 days of study drugs, and on isolates from patients with positive sputum cultures at the day 42 study visit to assess for the development of acquired drug resistance. Isolates will be tested against INH, rifampicin, pyrazinamide, ethambutol and the subject's assigned study drug. Patients who are found to be resistant to their assigned study drug at baseline will not be analyzable. After the initial treatment, all subjects will receive 6 months of standard TB treatment outside of the hospital.

ELIGIBILITY:
Inclusion Criteria:

-Adults, male or female, age 18 to 65 years. -Women with child-bearing potential (not surgically sterilized or postmenopausal for less than 1 year) must be using or agree to use an adequate method of birth control [condom; intravaginal spermicide (foams, jellies, sponge) and diaphragm; cervical cap or intrauterine device] during study drug treatment. -Newly diagnosed sputum smear-positive pulmonary tuberculosis as confirmed by sputum acid fast bacilli (AFB) smear and chest X-ray findings consistent with pulmonary tuberculosis. -Willing and able to provide informed consent. -Reasonably normal hemoglobin (greater than or equal to 8 gm/dL), renal function (serum creatinine less than 2 mg/dL), hepatic function [serum aspartate aminotransferase (AST) less than 1.5 times the upper limit of normal for the testing laboratory and total bilirubin less than 1.3 mg/dL], and random blood glucose less than 150 mg/dL.

Exclusion Criteria:

-Human immunodeficiency virus (HIV) infection. -Weight less than 75 percent of ideal body weight. -Presence of significant hemoptysis. Patients who cough up frank blood (more than blood streaked sputum) will not be eligible for enrollment. -Pregnant or breastfeeding women and those who are not practicing birth control. -Significant respiratory impairment (respiratory rate greater than 35/minute). -Clinical suspicion of disseminated tuberculosis or tuberculosis meningitis. -Presence of serious underlying medical illness, such as liver failure, renal failure, diabetes mellitus, chronic alcoholism, decompensated heart failure, hematologic malignancy or patients receiving myelosuppressive chemotherapy. -Patients receiving any of the following medications - monoamine oxidase inhibitors (phenelzine, tranylcypromine), adrenergic/serotonergic agonists such as pseudoephedrine and phenylpropanolamine (frequently found in cold and cough remedies), tricyclic antidepressants (amitriptyline, nortriptyline, protriptyline, doxepin, amoxapine, etc), antipsychotics such as chlorpromazine and buspirone, serotonin re-uptake inhibitors (fluoxetine, paroxetine, sertraline, etc.), buproprion, agents known to prolong the QTc interval [erythromycin, clarithromycin, astemizole, type Ia (quinidine, procainamide, disopyramide) and III (amiodarone, sotalol) anti-arrhythmics, carbamazepine, insulin, sulfonylureas, and meperidine. -Presence of QTc prolongation (greater than 450 msec) on baseline electrocardiogram (EKG). -Allergy or contraindication to use of study drugs. -Treatment with antituberculosis medications or other antibiotics with known activity against M. tuberculosis during the preceding 6 months. -Inability to provide informed consent. -Total white blood cell count less than 3000/mm^3. -Platelet count less than 150,000/mm^3. -Patients with suspected drug resistant tuberculosis (e.g., contact to source patient with drug resistant tuberculosis, patients who have relapsed after previous treatment for tuberculosis). -Patients likely, in the opinion of the local investigator, to be unable to comply with the requirements of the study protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2004-02-10 (Actual); Primary Completion 2007-11-23 (Actual); Study Completion 2007-12-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- San Francisco General Hospital - Pulmonary and Critical Care Medicine, San Francisco, California, United States
- Universidade Federal do Espirito Santo - Duke Hubert-Yeargan Center, Vitória, Espírito Santo, Brazil

REFERENCES:
- [Result] Johnson JL, Hadad DJ, Boom WH, Daley CL, Peloquin CA, Eisenach KD, Jankus DD, Debanne SM, Charlebois ED, Maciel E, Palaci M, Dietze R. Early and extended early bactericidal activity of levofloxacin, gatifloxacin and moxifloxacin in pulmonary tuberculosis. Int J Tuberc Lung Dis. 2006 Jun;10(6):605-12. PMID 16776446
- [Result] Dietze R, Hadad DJ, McGee B, Molino LP, Maciel EL, Peloquin CA, Johnson DF, Debanne SM, Eisenach K, Boom WH, Palaci M, Johnson JL. Early and extended early bactericidal activity of linezolid in pulmonary tuberculosis. Am J Respir Crit Care Med. 2008 Dec 1;178(11):1180-5. doi: 10.1164/rccm.200806-892OC. Epub 2008 Sep 11. PMID 18787216
- [Result] Millard J, Pertinez H, Bonnett L, Hodel EM, Dartois V, Johnson JL, Caws M, Tiberi S, Bolhuis M, Alffenaar JC, Davies G, Sloan DJ. Linezolid pharmacokinetics in MDR-TB: a systematic review, meta-analysis and Monte Carlo simulation. J Antimicrob Chemother. 2018 Jul 1;73(7):1755-1762. doi: 10.1093/jac/dky096. PMID 29584861
- [Result] Peloquin CA, Hadad DJ, Molino LP, Palaci M, Boom WH, Dietze R, Johnson JL. Population pharmacokinetics of levofloxacin, gatifloxacin, and moxifloxacin in adults with pulmonary tuberculosis. Antimicrob Agents Chemother. 2008 Mar;52(3):852-7. doi: 10.1128/AAC.01036-07. Epub 2007 Dec 10. PMID 18070980
- [Result] McGee B, Dietze R, Hadad DJ, Molino LP, Maciel EL, Boom WH, Palaci M, Johnson JL, Peloquin CA. Population pharmacokinetics of linezolid in adults with pulmonary tuberculosis. Antimicrob Agents Chemother. 2009 Sep;53(9):3981-4. doi: 10.1128/AAC.01378-08. Epub 2009 Jun 29. PMID 19564361
- [Result] Li L, Mahan CS, Palaci M, Horter L, Loeffelholz L, Johnson JL, Dietze R, Debanne SM, Joloba ML, Okwera A, Boom WH, Eisenach KD. Sputum Mycobacterium tuberculosis mRNA as a marker of bacteriologic clearance in response to antituberculosis therapy. J Clin Microbiol. 2010 Jan;48(1):46-51. doi: 10.1128/JCM.01526-09. Epub 2009 Nov 18. PMID 19923475

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening for the trial began in February 2004 in Vitória, Brazil. Non-HIV infected adults aged 18-65 years with suspected pulmonary tuberculosis (TB) were recruited at local TB posts and the Hospital Universitario Cassiano Antonio de Moraes of the Universidade Federal do Espírito Santo (UFES) in Vitória. Enrollment was completed in October 2007.
Pre-assignment Details: A total of 113 adults with suspected pulmonary TB were evaluated for study participation. Forty-three were excluded because they did not meet the eligibility criteria, leaving a total of 70 patients.
Groups:
- Gatifloxacin 400 mg/Day: Gatifloxacin 400 mg/day x 7 days
- Levofloxacin 1000 mg/Day: Levofloxacin 1000 mg/day x 7days
- Linezolid 600 mg / Once Daily: Linezolid 600 mg/once daily x 7days
- Linezolid 600 mg / Twice Daily: Linezolid 600 mg twice daily x 7 days
- Moxifloxacin 400 mg/Day: Moxifloxacin 400 mg/day x 7 days
- Isoniazid (INH) 300 mg/Day: Isoniazid (INH) 300 mg/day x 7 days
Period: Overall Study
Arm/Group | Gatifloxacin 400 mg/Day | Levofloxacin 1000 mg/Day | Linezolid 600 mg / Once Daily | Linezolid 600 mg / Twice Daily | Moxifloxacin 400 mg/Day | Isoniazid (INH) 300 mg/Day
Started | 10 | 10 | 10 | 10 | 10 | 20
Completed | 10 | 10 | 10 | 9 | 9 | 18
Not Completed | 0 | 0 | 0 | 1 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gatifloxacin 400 mg/Day | Levofloxacin 1000 mg/Day | Linezolid 600 mg / Once Daily | Linezolid 600 mg / Twice Daily | Moxifloxacin 400 mg/Day | Isoniazid (INH) 300 mg/Day | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 20 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 10 | 10 | 20 | 70
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34.5 (10.1) [27.0 to 40.0] | 43.5 (6.4) [42.0 to 46.0] | 33.5 (13.4) [23.0 to 42.0] | 45.0 (12.7) [39.0 to 48.0] | 35.0 (8.4) [25.0 to 37.0] | 33.0 (11.4) [23.0 to 43.5] | 35.0 (11.2) [26.0 to 44.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 2 | 1 | 3 | 11
  Male | 9 | 8 | 8 | 8 | 9 | 17 | 59
Region of Enrollment [Number; unit: participants]
  Brazil | 10 | 10 | 10 | 10 | 10 | 20 | 70

OUTCOME MEASURES:

1. Primary Outcome: Sputum Bacillary Loads: Adjusted Area Under the Curve (aAUC)
Description: The adjusted area under the curve (aAUC) for sputum colony forming units (cfu) for each day on treatment was calculated. The aAUC represents the percentage of the expected AUC given no change in log cfu in response to study drug administration.
Time Frame: Study drug administration duration - 7 days monotherapy
Population: The aAUC was calculated for 10 subjects per treatment arm (n=40).
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Gatifloxacin 400 mg/Day | Levofloxacin 1000 mg/Day | Moxifloxacin 400 mg/Day | Isoniazid (INH) 300 mg/Day
Number analyzed (Participants) | 10 | 10 | 10 | 10
Percentage
  Day 1 | 0.98 (0.03) | 0.98 (0.03) | 0.96 (0.04) | 0.95 (0.03)
  Day 2 | 0.96 (0.03) | 0.95 (0.05) | 0.94 (0.06) | 0.90 (0.04)
  Day 3 | 0.92 (0.05) | 0.91 (0.07) | 0.91 (0.08) | 0.87 (0.04)
  Day 4 | 0.89 (0.07) | 0.88 (0.08) | 0.89 (0.09) | 0.84 (0.04)
  Day 5 | 0.87 (0.08) | 0.85 (0.09) | 0.87 (0.10) | 0.81 (0.05)
  Day 6 | 0.85 (0.08) | 0.83 (0.10) | 0.85 (0.10) | 0.80 (0.06)
  Day 7 | 0.82 (0.09) | 0.81 (0.10) | 0.83 (0.10) | 0.80 (0.06)
Statistical Analysis 1: Comparison: Gatifloxacin 400 mg/Day vs Levofloxacin 1000 mg/Day vs Moxifloxacin 400 mg/Day vs Isoniazid (INH) 300 mg/Day; Mean adjusted aAUC for all 4 treatment groups over the 7 days of study drug administration; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Gatifloxacin 400 mg/Day vs Levofloxacin 1000 mg/Day vs Moxifloxacin 400 mg/Day vs Isoniazid (INH) 300 mg/Day; Day 1. Pooled sputum bacillary load data for patients in the 3 fluoroquinolones arms were combined and compared to that of patients in the INH arm; Test type: Superiority or Other; p = 0.041, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Gatifloxacin 400 mg/Day vs Levofloxacin 1000 mg/Day vs Moxifloxacin 400 mg/Day vs Isoniazid (INH) 300 mg/Day; Day 2. Pooled sputum bacillary load data for patients in the 3 fluoroquinolones arms were combined and compared to that of patients in the INH arm; Test type: Superiority or Other; p = 0.008, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Gatifloxacin 400 mg/Day vs Levofloxacin 1000 mg/Day vs Moxifloxacin 400 mg/Day vs Isoniazid (INH) 300 mg/Day; Day 3. Pooled sputum bacillary load data for patients in the 3 fluoroquinolones arms were combined and compared to that of patients in the INH arm; Test type: Superiority or Other; p = 0.012, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Gatifloxacin 400 mg/Day vs Levofloxacin 1000 mg/Day vs Moxifloxacin 400 mg/Day vs Isoniazid (INH) 300 mg/Day; Day 4. Pooled sputum bacillary load data for patients in the 3 fluoroquinolones arms were combined and compared to that of patients in the INH arm; Test type: Superiority or Other; p = 0.01, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Gatifloxacin 400 mg/Day vs Levofloxacin 1000 mg/Day vs Moxifloxacin 400 mg/Day vs Isoniazid (INH) 300 mg/Day; Day 5. Pooled sputum bacillary load data for patients in the 3 fluoroquinolones arms were combined and compared to that of patients in the INH arm; Test type: Superiority or Other; p = 0.03, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Gatifloxacin 400 mg/Day vs Levofloxacin 1000 mg/Day vs Moxifloxacin 400 mg/Day vs Isoniazid (INH) 300 mg/Day; Day 6. Pooled sputum bacillary load data for patients in the 3 fluoroquinolones arms were combined and compared to that of patients in the INH arm; Test type: Superiority or Other; p = 0.091, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Gatifloxacin 400 mg/Day vs Levofloxacin 1000 mg/Day vs Moxifloxacin 400 mg/Day vs Isoniazid (INH) 300 mg/Day; Day 7. Pooled sputum bacillary load data for patients in the 3 fluoroquinolones arms were combined and compared to that of patients in the INH arm; Test type: Superiority or Other; p = 0.354, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Sputum mRNA Clearance Rate - Results Are Pending.
Time Frame: Study drug administration duration
Reporting Status: Not Posted

3. Secondary Outcome: Sputum Cytokine Proteins - Results Are Pending.
Time Frame: Study drug administration duration
Reporting Status: Not Posted

4. Secondary Outcome: Maximum Plasma Drug Concentration (Cmax)
Description: Maximum plasma concentration, given sampling scheme
Time Frame: Day 5 (7 time points)
Population: Thirty-nine patients underwent pharmacokinetic (PK) sampling after receiving 5 daily doses of study drug. Plasma samples were collected at 7 time points on the 5th day after beginning study drug monotherapy. One subject in the moxifloxacin arm was discontinued from the study before day 5 and did not undergo PK sampling.
Measure: Median (Full Range); unit: ug/ml
Arm/Group | Gatifloxacin 400 mg/Day | Levofloxacin 1000 mg/Day | Moxifloxacin 400 mg/Day | Isoniazid (INH) 300 mg/Day
Number analyzed (Participants) | 10 | 10 | 9 | 10
ug/ml | 4.8 [3.8 to 6.4] | 15.6 [8.6 to 43.0] | 6.1 [4.5 to 9.0] | 3.6 [2.5 to 6.1]

5. Primary Outcome: Difference in Sputum Bacillary Loads: Early Bactericidal Activity (EBA) Days 0 to 2; Fluoroquinolones/Isoniazid (INH) Comparison
Description: Early bactericidal activity (EBA 0-2) was calculated as the rate of fall in sputum colony forming units (cfu) (expressed in log10 units) during the first 2 days of monotherapy.
Time Frame: Day 0 to Day 2 Monotherapy
Population: Early bactericidal activity (EBA 0-2) was calculated for 10 subjects per treatment arm (n=40).
Measure: Mean (Standard Deviation); unit: log10 cfu/ml/day
Arm/Group | Gatifloxacin 400 mg/Day | Levofloxacin 1000 mg/Day | Moxifloxacin 400 mg/Day | Isoniazid (INH) 300 mg/Day
Number analyzed (Participants) | 10 | 10 | 10 | 10
log10 cfu/ml/day | 0.35 (0.27) | 0.45 (0.35) | 0.33 (0.39) | 0.67 (0.17)
Statistical Analysis 1: Comparison: Gatifloxacin 400 mg/Day vs Levofloxacin 1000 mg/Day vs Moxifloxacin 400 mg/Day vs Isoniazid (INH) 300 mg/Day; Mean values of EBA Days 0 to 2 for the 4 treatment groups were compared; Test type: Superiority or Other; p = 0.05, ANOVA
Statistical Analysis 2: Comparison: Gatifloxacin 400 mg/Day vs Isoniazid (INH) 300 mg/Day; Two way comparison of INH against gatifloxacin using a simultaneous non-parametric procedure; Test type: Superiority or Other; p = 0.01, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Moxifloxacin 400 mg/Day vs Isoniazid (INH) 300 mg/Day; Two way comparison of INH against moxifloxacin using a simultaneous non-parametric procedure; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Levofloxacin 1000 mg/Day vs Isoniazid (INH) 300 mg/Day; Two way comparison of INH against levofloxacin using a simultaneous non-parametric procedure; Test type: Superiority or Other; p = 0.14, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Extended Early Bactericidal Activity (EBA) From Days 2 to 7; Fluoroquinolones/Isoniazid (INH) Comparison
Description: The rate of fall in sputum cfu between day 2 and day 7 of monotherapy was estimated by the slope of the linear regression obtained by fitting the 6 sputum cfu values corresponding to Days 2 through 7.
Time Frame: Day 2 to Day 7 Monotherapy
Population: A total of 38 patients were analyzed for Early Bactericidal Activity (EBA) Days 2-7. One patient in the moxifloxacin arm discontinued the study drug after 4 days. One patient in the INH arm discontinued the study drug after 6 days.
Measure: Mean (Standard Deviation); unit: log10 cfu/ml/day
Arm/Group | Gatifloxacin 400 mg/Day | Levofloxacin 1000 mg/Day | Moxifloxacin 400 mg/Day | Isoniazid (INH) 300 mg/Day
Number analyzed (Participants) | 10 | 10 | 9 | 9
log10 cfu/ml/day | 0.17 (0.13) | 0.18 (0.13) | 0.17 (0.09) | 0.08 (0.09)
Statistical Analysis 1: Comparison: Gatifloxacin 400 mg/Day vs Levofloxacin 1000 mg/Day vs Moxifloxacin 400 mg/Day vs Isoniazid (INH) 300 mg/Day; Mean values of EBA Days 2 to 7 for the 4 treatment groups were compared; Test type: Superiority or Other; p = 0.51, ANOVA
Statistical Analysis 2: Comparison: Gatifloxacin 400 mg/Day vs Levofloxacin 1000 mg/Day vs Moxifloxacin 400 mg/Day vs Isoniazid (INH) 300 mg/Day; The rate of fall in sputum cfu for the 4 treatment groups between day 2 and day 7 of monotherapy was estimated by the slope of the linear regression obtained from fitting the 6 sputum cfu values corresponding to days 2 through 7; Test type: Superiority or Other; p = 0.16, ANOVA
Statistical Analysis 3: Comparison: Gatifloxacin 400 mg/Day vs Levofloxacin 1000 mg/Day vs Moxifloxacin 400 mg/Day vs Isoniazid (INH) 300 mg/Day; EBA Days 2-7 for patients in the 3 fluoroquinolone groups were pooled and compared to bactericidal activity of patients in the INH arm; Test type: Superiority or Other; p = 0.036, Wilcoxon (Mann-Whitney)

7. Primary Outcome: Sputum Bacillary Loads: Adjusted Area Under the Curve (aAUC)
Description: The adjusted area under the curve (aAUC) for sputum colony forming unit (cfu) for each day on treatment was calculated for patients in the INH arm and those in the Linezolid once daily and Linezolid twice daily arms. The aAUC represents the percentage of the expected AUC given no change in log cfu in response to study drug administration.
Time Frame: Study drug administration duration - 7 days monotherapy
Population: The aAUC was calculated for 29 patients. One patient in the linezolid twice daily arm withdrew after randomization before receiving any doses of study drug.
Measure: Mean (Standard Deviation); unit: Percentage
Groups:
- Isoniazid 300 mg/Day: Isoniazid (INH) 300 mg/day x 7 days
- Linezolid 600 mg/Once Daily: Linezolid, 600 mg/day x 7 days
- Linezolid 600 mg/Twice Daily: Linezolid 600 mg q12h x 7 days
Arm/Group | Isoniazid 300 mg/Day | Linezolid 600 mg/Once Daily | Linezolid 600 mg/Twice Daily
Number analyzed (Participants) | 10 | 10 | 9
Percentage
  Day 1 | 0.94 (0.06) | 0.98 (0.04) | 0.98 (0.04)
  Day 2 | 0.89 (0.08) | 0.97 (0.07) | 0.96 (0.07)
  Day 3 | 0.89 (0.03) | 0.96 (0.07) | 0.95 (0.08)
  Day 4 | 0.85 (0.09) | 0.96 (0.07) | 0.94 (0.08)
  Day 5 | 0.83 (0.10) | 0.95 (0.07) | 0.94 (0.08)
  Day 6 | 0.81 (0.12) | 0.95 (0.07) | 0.93 (0.07)
  Day 7 | 0.83 (0.07) | 0.95 (0.07) | 0.93 (0.07)
Statistical Analysis 1: Comparison: Isoniazid 300 mg/Day vs Linezolid 600 mg/Once Daily vs Linezolid 600 mg/Twice Daily; Mean adjusted aAUC for all 3 treatment groups over the 7 days of study drug administration; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Isoniazid 300 mg/Day vs Linezolid 600 mg/Once Daily vs Linezolid 600 mg/Twice Daily; Day 1. Pooled sputum bacillary load data for patients in the linezolid arms were combined and compared to that of patients in the INH arm; Test type: Superiority or Other; p = 0.023, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Isoniazid 300 mg/Day vs Linezolid 600 mg/Once Daily vs Linezolid 600 mg/Twice Daily; Day 2. Pooled sputum bacillary load data for patients in the linezolid arms were combined and compared to that of patients in the INH arm; Test type: Superiority or Other; p = 0.018, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Isoniazid 300 mg/Day vs Linezolid 600 mg/Once Daily vs Linezolid 600 mg/Twice Daily; Day 3. Pooled sputum bacillary load data for patients in the linezolid arms were combined and compared to that of patients in the INH arm; Test type: Superiority or Other; p = 0.03, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Isoniazid 300 mg/Day vs Linezolid 600 mg/Once Daily vs Linezolid 600 mg/Twice Daily; Day 4. Pooled sputum bacillary load data for patients in the linezolid arms were combined and compared to that of patients in the INH arm; Test type: Superiority or Other; p = 0.012, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Isoniazid 300 mg/Day vs Linezolid 600 mg/Once Daily vs Linezolid 600 mg/Twice Daily; Day 5. Pooled sputum bacillary load data for patients in the linezolid arms were combined and compared to that of patients in the INH arm; Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Isoniazid 300 mg/Day vs Linezolid 600 mg/Once Daily vs Linezolid 600 mg/Twice Daily; Day 6. Pooled sputum bacillary load data for patients in the linezolid arms were combined and compared to that of patients in the INH arm; Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Isoniazid 300 mg/Day vs Linezolid 600 mg/Once Daily vs Linezolid 600 mg/Twice Daily; Day 7. Pooled sputum bacillary load data for patients in the linezolid arms were combined and compared to that of patients in the INH arm; Test type: Superiority or Other; p = 0.004, Wilcoxon (Mann-Whitney)

8. Primary Outcome: Difference in Sputum Bacillary Loads: Early Bactericidal Activity (EBA) Days 0 to 2; Linezolid Once Daily/Linezolid Twice Daily/Isoniazid (INH) Comparison
Description: Early bactericidal activity (EBA 0-2) was calculated as the rate of fall in sputum cfu (expressed in log10 units) during the first 2 days of monotherapy. Mean values for the 3 treatment groups were compared.
Time Frame: Day 0 to Day 2 Monotherapy
Population: EBA 0-2 comparisons across groups were done for 29 patients. One patient in the linezolid twice daily arm withdrew from the study after randomization before receiving any doses of study drug.
Measure: Mean (Standard Deviation); unit: log10 cfu/ml/day
Arm/Group | Isoniazid 300 mg/Day | Linezolid 600 mg/Once Daily | Linezolid 600 mg/Twice Daily
Number analyzed (Participants) | 10 | 10 | 9
log10 cfu/ml/day | 0.67 (0.35) | 0.18 (0.27) | 0.26 (0.42)
Statistical Analysis 1: Comparison: Isoniazid 300 mg/Day vs Linezolid 600 mg/Once Daily vs Linezolid 600 mg/Twice Daily; Mean values of EBA Days 0 to 2 for the 3 treatments groups were compared; Test type: Superiority or Other; p < 0.01, ANOVA
Statistical Analysis 2: Comparison: Isoniazid 300 mg/Day vs Linezolid 600 mg/Once Daily; Two way comparison of INH against Linezolid once daily using a simultaneous non-parametric procedure; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Isoniazid 300 mg/Day vs Linezolid 600 mg/Once Daily vs Linezolid 600 mg/Twice Daily; Mean EBA 0-2 of INH was compared to pooled Linezolid once daily and Linezolid twice daily results; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Time to Maximum Plasma Drug Concentration (Tmax) and Half-life
Time Frame: Day 5 (7 time points)
Population: Thirty-nine patients underwent pharmacokinetic (PK) sampling after receiving 5 daily doses of study drug. One subject in the moxifloxacin arm was discontinued from the study before day 5 and did not undergo PK sampling.
Measure: Median (Full Range); unit: hours
Arm/Group | Gatifloxacin 400 mg/Day | Levofloxacin 1000 mg/Day | Moxifloxacin 400 mg/Day | Isoniazid (INH) 300 mg/Day
Number analyzed (Participants) | 10 | 10 | 9 | 10
hours
  Tmax | 1.5 [1.0 to 8.0] | 1.0 [1.0 to 4.0] | 1.0 [1.0 to 2.0] | 1 [1.0 to 2.0]
  Half-life | 6.0 [5.2 to 9.3] | 7.6 [4.4 to 19.1] | 8.1 [5.1 to 9.9] | 2.5 [1.5 to 4.9]

10. Secondary Outcome: Maximum Plasma Drug Concentration/Minimum Inhibitory Concentration (Cmax/MIC)
Time Frame: Day 5 (7 time points)
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: ug/ml
Groups:
- Levofloxacin 1000 mg/Day: Levofloxacin 1000 mg/day x 7 days
Arm/Group | Gatifloxacin 400 mg/Day | Levofloxacin 1000 mg/Day | Moxifloxacin 400 mg/Day | Isoniazid (INH) 300 mg/Day
Number analyzed (Participants) | 10 | 10 | 9 | 10
ug/ml | 9.5 [8.4 to 11.3] | 15.6 [12.2 to 16.6] | 12.3 [9.6 to 13.4] | 70.6 [64.0 to 76.2]

11. Primary Outcome: Difference in Sputum Bacillary Loads: Extended Early Bactericidal Activity (EBA) From Days 2 to 7; Linezolid Once Daily/Linezolid Twice Daily/INH Comparison
Description: as for outcome 6
Time Frame: Day 2 to Day 7 Monotherapy
Population: One patient in the INH arm discontinued the study drug after 5 days. Days 3 and 7 cultures for another patient in the INH arm were contaminated and cfu data are not available for this patient. One patient in the linezolid twice daily arm withdrew from the study after randomization before receiving any doses of study drug.
Measure: Mean (Standard Deviation); unit: log10 cfu/ml
Arm/Group | Isoniazid 300 mg/Day | Linezolid 600 mg/Once Daily | Linezolid 600 mg/Twice Daily
Number analyzed (Participants) | 8 | 10 | 9
log10 cfu/ml | 0.16 (0.11) | 0.09 (0.17) | 0.04 (0.11)
Statistical Analysis 1: Comparison: Isoniazid 300 mg/Day vs Linezolid 600 mg/Once Daily vs Linezolid 600 mg/Twice Daily; Mean values EBA Days 2-7 for the 3 treatment groups were compared; Test type: Superiority or Other; p = 0.25, ANOVA
Statistical Analysis 2: Comparison: Isoniazid 300 mg/Day vs Linezolid 600 mg/Once Daily vs Linezolid 600 mg/Twice Daily; The rate of fall in sputum cfu for the 3 treatment groups between day 2 and day 7 of monotherapy was estimated by the slope of the linear regression obtained from fitting the 6 sputum cfu values corresponding to days 2 through 7; Test type: Superiority or Other; p = 0.42, ANOVA
Statistical Analysis 3: Comparison: Isoniazid 300 mg/Day vs Linezolid 600 mg/Once Daily vs Linezolid 600 mg/Twice Daily; EBA Days 2-7 for INH was compared to that of the pooled linezolid arms; Test type: Superiority or Other; p = 0.14, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Pharmacokinetic Parameters: Area Under the Curve (AUC) During First 12 and 24 Hours
Description: Area under the curve (AUC), from time 0-12 hours for INH or 0-24 hours for gatifloxacin, levofloxacin, and moxifloxacin.
Time Frame: Day 5 (7 time points)
Population: as for outcome 4
Measure: Median (Full Range); unit: ug/h/ml
Arm/Group | Gatifloxacin 400 mg/Day | Levofloxacin 1000 mg/Day | Moxifloxacin 400 mg/Day | Isoniazid (INH) 300 mg/Day
Number analyzed (Participants) | 10 | 10 | 9 | 10
ug/h/ml | 42.8 [31.7 to 51.0] | 129.1 [103.4 to 358.3] | 55.3 [36.0 to 79.1] | 11.9 [7.1 to 37.4]

13. Secondary Outcome: Area Under the Curve During First 12 or 24 Hours / Minimum Inhibitory Concentration (AUC/MIC)
Description: Area Under the Curve (AUC) During First 12 or 24 Hours /Minimum Inhibitory Concentration. AUC reflects total drug (bound and unbound). MIC values were determined using protein-containing media.
Time Frame: Day 5 (7 time points)
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: ug/ml
Arm/Group | Gatifloxacin 400 mg/Day | Levofloxacin 1000 mg/Day | Moxifloxacin 400 mg/Day | Isoniazid (INH) 300 mg/Day
Number analyzed (Participants) | 10 | 10 | 9 | 10
ug/ml | 85.6 [70.7 to 89.7] | 129.1 [121.0 to 145.0] | 110.5 [98.9 to 121.6] | 215.2 [177.4 to 329.6]

14. Secondary Outcome: Maximum Plasma Drug Concentration (Cmax)
Description: Maximum Plasma Drug Concentration (Cmax), given sampling scheme
Time Frame: Day 5 (7 time points)
Population: Twenty-nine patients underwent pharmacokinetic (PK) sampling after receiving 5 daily doses of study drug. One subject in the linezolid twice daily arm withdrew from the study after randomization before receiving any doses of study drug.
Measure: Median (Full Range); unit: ug/ml
Arm/Group | Isoniazid 300 mg/Day | Linezolid 600 mg/Once Daily | Linezolid 600 mg/Twice Daily
Number analyzed (Participants) | 10 | 10 | 9
ug/ml | 3.3 [2.5 to 5.3] | 15.0 [11.9 to 21.3] | 19.4 [11.8 to 24.9]

15. Secondary Outcome: Time to Maximum Plasma Drug Concentration (Tmax) and Half-life
Time Frame: Day 5 (7 time points)
Population: as for outcome 14
Measure: Median (Full Range); unit: hours
Arm/Group | Isoniazid 300 mg/Day | Linezolid 600 mg/Once Daily | Linezolid 600 mg/Twice Daily
Number analyzed (Participants) | 10 | 10 | 9
hours
  Tmax in h (apparent time of max plasma conc.) | 1.0 [1.0 to 2.0] | 1.5 [1.0 to 4.0] | 1.0 [1.0 to 4.0]
  Half-life | 3.6 [1.1 to 4.5] | 3.20 [1.5 to 5.0] | 4.56 [2.1 to 7.0]

16. Secondary Outcome: Pharmacokinetic Parameters: Area Under the Curve During First 12 and 24 Hours
Description: Median pharmacokinetic parameters (range). AUC 0-12 and AUC 0-24 = area under the curve during the first 12 and 24 hours after dosing, respectively
Time Frame: Day 5 (7 time points)
Population: as for outcome 14
Measure: Median (Full Range); unit: ug/h/ml
Arm/Group | Isoniazid 300 mg/Day | Linezolid 600 mg/Once Daily | Linezolid 600 mg/Twice Daily
Number analyzed (Participants) | 10 | 10 | 9
ug/h/ml
  AUC 0-12 (ug/h/ml) | 17.0 [6.5 to 26.9] | 87.0 [47.5 to 119.3] | 116.4 [50.4 to 197.2]
  AUC 0-24 (ug/h/ml) | 19.2 [6.5 to 29.0] | 96.9 [47.8 to 143.7] | 232.9 [100.8 to 394.4]

17. Secondary Outcome: Maximum Plasma Drug Concentrations (Cmax), Adjusted for Free Drug Concentration
Description: Cmax adjusted for free drug concentrations after 5 days of monotherapy with study drugs
Time Frame: Day 5 (7 time points)
Population: as for outcome 14
Measure: Median (Full Range); unit: ug/ml
Arm/Group | Isoniazid 300 mg/Day | Linezolid 600 mg/Once Daily | Linezolid 600 mg/Twice Daily
Number analyzed (Participants) | 10 | 10 | 9
ug/ml | 3.1 [2.5 to 4.8] | 10.3 [8.2 to 14.7] | 13.4 [8.1 to 17.2]

18. Secondary Outcome: Maximum Plasma Drug Concentration/Minimum Inhibitory Concentration (Cmax/MIC) Adjusted for Free Drug Concentrations
Time Frame: Day 5 (7 time points)
Population: Twenty-nine patients underwent pharmacodynamic sampling after receiving 5 daily doses of study drug. One subject in the linezolid twice daily arm withdrew from the study after randomization before receiving any doses of study drug.
Measure: Median (Inter-Quartile Range); unit: ug/ml
Arm/Group | Isoniazid 300 mg/Day | Linezolid 600 mg/Once Daily | Linezolid 600 mg/Twice Daily
Number analyzed (Participants) | 10 | 10 | 9
ug/ml | 62.7 [51.0 to 77.3] | 20.0 [10.2 to 21.9] | 16.2 [14.3 to 23.0]

19. Secondary Outcome: Area Under the Curve (AUC) During First 12 and 24 Hours Adjusted for Free Drug Concentrations
Description: Median pharmacodynamic parameters (range) adjusted for free drug concentrations. AUC 0-12 and AUC 0-24 = area under the curve during the first 12 and 24 hours after dosing, respectively
Time Frame: Day 5 (7 time points)
Population: Twenty-nine patients underwent pharmacodynamic (PD) sampling after receiving 5 daily doses of study drug. One subject in the linezolid twice daily arm withdrew from the study after randomization before receiving any doses of study drug.
Measure: Median (Inter-Quartile Range); unit: ug/h/ml
Arm/Group | Isoniazid 300 mg/Day | Linezolid 600 mg/Once Daily | Linezolid 600 mg/Twice Daily
Number analyzed (Participants) | 10 | 10 | 9
ug/h/ml
  AUC 0-12 | 15.3 [5.8 to 24.2] | 60.1 [32.8 to 82.3] | 80.3 [34.8 to 136.1]
  AUC 0-24 | 17.2 [5.8 to 26.1] | 66.8 [33.0 to 99.2] | 160.7 [134.4 to 225.8]

20. Secondary Outcome: Area Under the Curve (AUC) Adjusted for Free Drug Concentrations/Minimum Inhibitory Concentration (MIC)
Description: Area Under the Curve 0-12 (AUC 0-12) Adjusted for Free Drug Concentrations/Minimum Inhibitory Concentration (MIC) and AUC 0-24/MIC
Time Frame: Day 5 (7 time points)
Population: as for outcome 19
Measure: Median (Inter-Quartile Range); unit: ug/h/ml
Arm/Group | Isoniazid 300 mg/Day | Linezolid 600 mg/Once Daily | Linezolid 600 mg/Twice Daily
Number analyzed (Participants) | 10 | 10 | 9
ug/h/ml
  AUC 0-12/MIC | 306.7 [229.3 to 405.2] | 107.8 [63.4 to 126.3] | 121.6 [79.8 to 141.6]
  AUC 0-24/MIC | 344.6 [249.4 to 449.2] | 116.2 [71.0 to 138.4] | 243.2 [159.7 to 283.2]

21. Secondary Outcome: Percent Dosing Interval Above Minimum Inhibitory Concentration (MIC)
Description: Determined by linear extrapolation of concentration-versus-time curve to intersection with MIC.
Time Frame: Day 5 (7 time points)
Population: as for outcome 19
Measure: Mean (Inter-Quartile Range); unit: Percentage
Groups:
- Linezolid 600 mg/Once Daily: Linezolid 600 mg/day x 7 days
Arm/Group | Isoniazid (INH) 300 mg/Day | Linezolid 600 mg/Once Daily | Linezolid 600 mg/Twice Daily
Number analyzed (Participants) | 10 | 10 | 10
Percentage | 95.5 [76.4 to 100] | 62.8 [54.6 to 77.0] | 100.0 [100 to 100]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from February 2004 through October 2007.
Description: Patients reported adverse events at scheduled or unscheduled visits. Adverse event forms were completed by medical officers on site.
Arm/Group | Gatifloxacin 400 mg/Day | Levofloxacin 1000 mg/Day | Linezolid 600 mg / Once Daily | Linezolid 600 mg / Twice Daily | Moxifloxacin 400 mg/Day | Isoniazid (INH) 300 mg/Day
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/20
Other Adverse Events (participants affected / at risk) | 8/10 | 7/10 | 8/10 | 5/10 | 7/10 | 7/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gatifloxacin 400 mg/Day (N=10) | Levofloxacin 1000 mg/Day (N=10) | Linezolid 600 mg / Once Daily (N=10) | Linezolid 600 mg / Twice Daily (N=10) | Moxifloxacin 400 mg/Day (N=10) | Isoniazid (INH) 300 mg/Day (N=20)
Acne (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 0 (0)
Elevated Monocytes (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematocrit Decreased (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin Decreased (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Intestinal Ancyclostomiasis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Intestinal Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Intestinal Strongyloidiasis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Joint Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lumbar Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in Both Shoulders (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Rales (or Crackles) (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (6) | 0 (0) | 0 (0) | 6 (13) | 7 (17)
Ronchi (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Sweating (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The small sample size had limited power to detect small differences in EBA between study arms even though we enrolled patients with smear-positive TB and high sputum bacillary burden to improve chances of detecting differences between treatment arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No